CLINICAL TRIAL: NCT06624176
Title: The Effect of ShotBlocker on Pain in Full Term Infants Undergoing Intramuscular Injection: A Randomized Controlled Trial
Brief Title: ShotBlocker During Intramuscular Injection Randomized Control Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lauren Fortier (Other)
Responsible Party: Sponsor-Investigator, Lauren Fortier, Instructor, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00001110
Record Dates: First submitted 2024-05-02; First posted 2024-10-02 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-09

CONDITIONS: Neonatal Pain
Keywords: ShotBlocker; Neonatal Pain; Needlestick
MeSH Terms: conditions — Needlestick Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- ShotBlocker Administration (Experimental): The treatment group will employ the medical device of interest, ShotBlocker, bundled with the standard-of-care comfort measures of swaddling and sucrose during the administration of the Hepatitis B Immunization. A Masimo Rad-97 Oximeter probe will be applied to record a baseline and intervention physiologic response. There will be an Opt-In Video Recording option to assign a pain score (PIPP Scale) during the procedure by a blinded medical professional.
  Interventions: Device: Bionix ShotBlocker; Other: Swaddling; Other: Sucrose administration; Other: Masimo Rad-97 Oximeter probe
- Standard of Care Comfort Tools (Active Comparator): The control group will employ the standard-of-care comfort measures of swaddling and sucrose during the administration of the Hepatitis B Immunization. A Masimo Rad-97 Oximeter probe will be applied to record a baseline and intervention physiologic response. There will be an Opt-In Video Recording option to assign a pain score (PIPP Scale) during the procedure by a blinded medical professional.
  Interventions: Other: Swaddling; Other: Sucrose administration; Other: Masimo Rad-97 Oximeter probe

INTERVENTIONS:
Device: Bionix ShotBlocker — This is a hospital-approved device used as standard-of-care in older children and adults to reduce pain during painful procedures. It is not considered established standard-of-care in the infant cohort.
  Arms: ShotBlocker Administration
Other: Swaddling — Standard of care swaddling
Other: Sucrose administration — Standard of care sucrose administration
Other: Masimo Rad-97 Oximeter probe — Oximeter probe

SUMMARY:
The objective of this trial is to evaluate the effect of Bionix ShotBlocker on pain of injection of the first Hepatitis B vaccine in healthy newborns. ShotBlocker is a pain reducing tool used in babies, children, and adults for injections. Swaddling during the injection and administration of oral sucrose prior to the injection are established standards of care for painful procedures in neonates. The investigators hypothesize that the use of ShotBlocker in addition to swaddling and oral sucrose administration will lessen the pain response.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at UMass Memorial Medical Center (UMMMC) via vaginal delivery or cesarean delivery and under the care of the nursery team
* Term infants (37 to 42 weeks gestational age)
* No acute illness that causes pain
* Apgar score above 7 at 5 minutes
* Have successfully attempted at least one oral feeding
* No circumcision in the last 6 hours
* Parental consent for Hepatitis B vaccine

Exclusion Criteria:

* Swallow dysfunction
* Congenital or genetic abnormalities
* Infants who were exposed to sedatives within the last 12 hours
* Infants with skin on thigh, hand, or foot that is not intact
* Diagnosis of Neonatal Abstinence Syndrome (NAS)
* Infants who are simultaneously receiving Hepatitis B Immunoglobulin or Nirsevimab (RSV vaccine)
* Department of Children and Families (DCF) custody

Ages: 37 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Difference in the heart rate before, during, and after Hepatitis B vaccine injection between the control and intervention groups. | up to 4 minutes
  The primary outcome measure is the difference in the physiologic response before, during, and after the injection between the control and intervention groups as reflected as heart rate. Difference in heart rate will be evaluated through the measurements of heart rate recorded by a Masimo Rad-97 Oximeter.
Difference in the blood oxygen saturation before, during, and after Hepatitis B vaccine injection between the control and intervention groups. | up to 4 minutes
  The primary outcome measure is the difference in the physiologic response before, during, and after the injection between the control and intervention groups as reflected by blood oxygen saturation. Difference in blood oxygen saturation will be evaluated through transcutaneous measurements recorded by a Masimo Rad-97 Oximeter.

SECONDARY OUTCOMES:
Difference in pain score before, during, and after Hepatitis B vaccine injection between the control and intervention groups. | up to 3 minutes
  The secondary outcome measure is the difference in the pain score using the Premature Infant Pain Profile (PIPP) before, during, and after injection between the control and intervention groups. PIPP scores range from 0 to 15 and a lower score indicates a better outcome. For example, a PIPP score of 0 indicates no pain. There will be an Opt-In Video Recording option to assign a PIPP score before, during, and after vaccine administration. Infant response will be filmed during injection and evaluated by a blinded medical professional that did not participate in study procedures to assign a PIPP score.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Fortier, CPNP, MSN, Principal Investigator — Pediatric Nurse Practitioner for the Department of Pediatrics & PICU
Locations (1):
- UMass Memorial Medical Center- Memorial Campus, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Talebi M, Amiri SRJ, Roshan PA, Zabihi A, Zahedpasha Y, Chehrazi M. The effect of concurrent use of swaddle and sucrose on the intensity of pain during venous blood sampling in neonate: a clinical trial study. BMC Pediatr. 2022 May 10;22(1):263. doi: 10.1186/s12887-022-03323-0. PMID 35538448
- [Background] Caglar S, Buyukyilmaz F, Cosansu G, Caglayan S. Effectiveness of ShotBlocker for Immunization Pain in Full-Term Neonates: A Randomized Controlled Trial. J Perinat Neonatal Nurs. 2017 Apr/Jun;31(2):166-171. doi: 10.1097/JPN.0000000000000256. PMID 28437308
- [Background] Drago LA, Singh SB, Douglass-Bright A, Yiadom MY, Baumann BM. Efficacy of ShotBlocker in reducing pediatric pain associated with intramuscular injections. Am J Emerg Med. 2009 Jun;27(5):536-43. doi: 10.1016/j.ajem.2008.04.011. PMID 19497458
- [Background] Susilawati, Susilawati, Soetjiningsih Soetjiningsih, Bagus Ngurah Putu Arhana and Ida Bagus Subanada. "Effectiveness of PainAway® on hepatitis B intramuscular injection in term neonates: a randomized controlled trial." Paediatrica Indonesiana 50 (2010): 214. doi:10.14238/PI50.4.2010.214-9
- [Background] McNair C, Campbell-Yeo M, Johnston C, Taddio A. Nonpharmacologic Management of Pain During Common Needle Puncture Procedures in Infants: Current Research Evidence and Practical Considerations: An Update. Clin Perinatol. 2019 Dec;46(4):709-730. doi: 10.1016/j.clp.2019.08.006. Epub 2019 Aug 26. PMID 31653304